CLINICAL TRIAL: NCT05989646
Title: Brain Activity Among Children With Overactive Bladder and Daytime Urinary Incontinence and Healthy Children, and Modulation of Brain Activity by Transcutaneous Electrical Nerve Stimulation - a Functional Magnetic Resonance Imaging Study
Brief Title: Brain Activity Among Children With Overactive Bladder and Daytime Urinary Incontinence and Healthy Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aalborg University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Regional Hospital West Jutland (Other); Regionshospital Nordjylland (Other Government)
Responsible Party: Principal Investigator, Kristina Thorsteinsson, Principal Investigator, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N-20210004
Record Dates: First submitted 2023-05-31; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Urinary Incontinence; Daytime Wetting; Urination Disorders; Urination Involuntary; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Manifestations; Behavioral Symptoms; Mental Disorders; Elimination Disorders
Keywords: Transcutaneous Electrical Nerve Stimulation; TENS; Functional Magnetic Resonance Imaging; fMRI
MeSH Terms: conditions — Urinary Incontinence; Diurnal Enuresis; Urination Disorders; Nocturnal Enuresis; Urologic Diseases; Lower Urinary Tract Symptoms; Urological Manifestations; Behavioral Symptoms; Mental Disorders; Elimination Disorders

STUDY DESIGN:
Intervention Model Description: Cross-sectional and interventional cohort study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transcutaneous Electric Nerve Stimulation (TENS) (Experimental): Sacral TENS
  Interventions: Device: Sacral TENS

INTERVENTIONS:
Device: Sacral TENS — Sacral TENS applied two hours daily for 10 weeks
  Other Names: Urotherapy

SUMMARY:
The aim of this study is to investigate whether the activity in brain areas controlling the bladder is different among children suffering from Overactive Bladder (OAB) and Daytime Urinary Incontinence (DUI) compared to age- and gender-matched healthy children without bladder symptoms. Moreover, the aim is to investigate if sacral transcutaneous electric nerve stimulation (TENS) has a central mechanism of action. Children with OAB and DUI will be recruited from involved pediatric departments, and functional magnetic resonance imaging (fMRI) will be performed before and after 10 weeks of sacral TENS. In healthy children without bladder symptoms, only the baseline fMRI will be performed.

DETAILED DESCRIPTION:
Daytime Urinary Incontinence (DUI) is a common condition among children affecting 2.1-21.8 % of children aged 4.5-17 years. DUI is most often caused by a functional overactive bladder (OAB) leading to urgent desire to void (urgency) and frequent urinations (frequency). In some children with functional OAB and DUI, the bladder detrusor is overactive when performing a urodynamic investigation, but this is not evident for all children suffering from OAB and DUI. The etiology of OAB and DUI is not yet fully established and might be multifactorial.

A few studies among adults have shown that adult women with OAB and DUI has more activity in brain areas controlling the bladder compared to adult women without bladder symptoms. Moreover, one study among adult women has shown a decrease in brain activity in areas controlling the bladder after sacral TENS treatment. This has led to a hypothesis that increased activity in the brain is a pathophysiological mechanism of OAB and DUI. Brain activity among children with OAB and DUI has not yet been investigated.

Therefore, the objectives of this study is:

1. To investigate the activity in brain areas controlling the bladder among children with OAB and DUI and age- and gender-matched children without bladder symptoms AND
2. To investigate if sacral TENS has a centrally modulatory effect on the brain activity in areas controlling the bladder among children with OAB and DUI.

Methods: The study consists of two sub-studies. The first sub-study is a cross-sectional study, whereas the second sub-study is an interventional cohort study. Forty-five children with OAB and DUI and 20 healthy children without bladder symptoms will be recruited. The study includes one structural MRI as well as two sessions of functional MRIs (only one functional MRI for healthy participants), one session prior to and after 10 weeks of sacral TENS treatment. The functional MRI session consist of a functional MRI with full bladder followed by a functional MRI with empty bladder. Moreover, the study participants and/or their parents are asked to fill in frequency and volume charts, Dry Pie, screening tools to rule out attention deficit hyperactivity disorder and autism spectrum disorders, and quality of life-questionnaires (WHO-5 and PinQ).

ELIGIBILITY:
Inclusion Criteria:

* Overactive Bladder as per International Children's Continence Society criteria (cases only).
* At least 2 incontinence episodes per week (cases only).
* No urinary tract symptoms (healthy participants only).
* More than 3 daily urinations.
* Normal clinical examination.

Exclusion Criteria:

* Known urogenital abnormality affecting the lower urinary tract function.
* Prior surgery in the urinary tract (except circumcision).
* Known neurological diseases or prior cerebral surgery.
* Known neuropsychiatric disorders or suspicion of those by screening.
* Treatment with pharmacological agents affecting the brain function.
* Prior treatment with Enuresis Alarm or Transcutaneous Electrical Nerve Stimulation.
* Prior or current treatment with mirabegron or oxybutynin.
* Current urinary tract infection.
* Current constipation according to Rome IV-criteria or faecal incontinence.
* Claustrophobia.
* Metallic items in the body contraindicating MRI-scans.
* Abnormal uroflowmetry (healthy participants only).

Ages: 6 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 65 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-04 (Estimated)

PRIMARY OUTCOMES:
Activity in brain areas controlling the bladder | Baseline
  Blood Oxygen Level Dependent (BOLD)-signals on functional MRIs, compared between children with Overactive Bladder and Daytime Urinary Incontinence and children without bladder symptoms.
Change in activity in brain areas controlling the bladder after TENS-treatment | Baseline AND immediately after the intervention
  Blood Oxygen Level Dependent (BOLD)-signals on functional MRIs, compared between responders and non-responders to TENS-treatment.

SECONDARY OUTCOMES:
Structural differences on MRI among children with OAB and DUI and healthy children | Baseline
  Volume of brain areas involved in bladder control (e.g. lateral nuclei in pons, prefrontal cortex, anterior cingulate cortex (ACC), insula, periaqueductal grey (PAG), the pontine micturition center (PMC), and hypothalamus)
Differences in Quality of Life (QoL) between children with OAB and DUI and healthy children | Baseline
  Assessment of QoL using WHO-5 among children with OAB and DUI and compare to QoL among children without bladder symptoms.
Change in WHO-5 score among children with OAB and DUI at baseline and after the intervention. | Baseline AND immediately after the intervention
  Assessment of QoL using WHO-5 among children with OAB and DUI prior to and after ten weeks of sacral TENS-treatment. WHO-5 (World Health Organization Quality of Life Brief Version) is a validated tool, assessing QoL as a total percent-score (range 0-100). A high score indicates better QoL.
Change in PinQ score among children with OAB and DUI at baseline and after the intervention. | Baseline AND immediately after the intervention
  Assessment of QoL using PinQ among children with OAB and DUI prior to and after ten weeks of sacral TENS treatment. PinQ (Pediatric Incontinence Questionnaire) is a validated tool, assessing QoL as a total score (range 0-80). A lower score indicates better QoL.
Change in WHO-5 score among children with OAB and DUI compared among responders and non-responders to sacral TENS treatment. | Immediately after the intervention
  Assessment of QoL using WHO-5 and compare among responders and non-responders to sacral TENS-treatment. WHO-5 (World Health Organization Quality of Life Brief Version) is a validated tool, assessing QoL as a total percent-score (range 0-100). A high score indicates better QoL.
Change in PinQ score among children with OAB and DUI compared among responders and non-responders to sacral TENS treatment. | Immediately after the intervention
  Assessment of QoL using PinQ and compare among responders and non-responders to sacral TENS-treatment. PinQ (Pediatric Incontinence Questionnaire) is a validated tool, assessing QoL as a total score (range 0-80). A lower score indicates better QoL.
Differences in maximum voided volume among responders and non-responders to sacral TENS treatment | Baseline AND immediately after the intervention
  Differences in maximum voided volume (MVV) in milliliters as assessed by the frequency and volume chart, compared among responders and non-responders to sacral TENS treatment.
Differences in voiding frequency among responders and non-responders to sacral TENS treatment | Baseline AND immediately after the intervention
  Differences in voiding frequency as assessed by the frequency and volume chart, compared among responders and non-responders to sacral TENS treatment.
Differences in VAS Urgency among responders and non-responders to sacral TENS treatment | Baseline AND immediately after the intervention
  Differences in VAS Urgency (visual analogue scale for urgency) in percent with a higher percent indicating a higher degree of urgency, compared among responders and non-responders to sacral TENS treatment.
Differences in urinary incontinence severity scores among responders and non-responders to sacral TENS treatment | Baseline AND immediately after the intervention
  Differences in urinary incontinence severity scores as assessed by Dry Pie, compared among responders and non-responders to sacral TENS treatment.

CONTACTS AND LOCATIONS:
Locations (4):
- Denmark (4):
  - Department of Pediatrics, Aalborg University Hospital, Aalborg
  - Department of Pediatrics, Aarhus University Hospital, Aarhus
  - Department of Pediatrics, Regional Hospital West Jutland, Herning
  - Department of Pediatrics, North Denmark Regional Hospital, Hjørring

REFERENCES:
- [Background] Warner TC, Baandrup U, Jacobsen R, Boggild H, Aunsholt Ostergaard PS, Hagstrom S. Prevalence of nocturia and fecal and urinary incontinence and the association to childhood obesity: a study of 6803 Danish school children. J Pediatr Urol. 2019 May;15(3):225.e1-225.e8. doi: 10.1016/j.jpurol.2019.02.004. Epub 2019 Feb 15. PMID 30930018
- [Background] von Gontard A, Overs C, Moritz AM, Thome-Granz S, Hussong J. Incontinence and headache in preschool children. Neurourol Urodyn. 2019 Nov;38(8):2280-2287. doi: 10.1002/nau.24134. Epub 2019 Aug 8. PMID 31397011
- [Background] Gur E, Turhan P, Can G, Akkus S, Sever L, Guzeloz S, Cifcili S, Arvas A. Enuresis: prevalence, risk factors and urinary pathology among school children in Istanbul, Turkey. Pediatr Int. 2004 Feb;46(1):58-63. doi: 10.1111/j.1442-200X.2004.01824.x. PMID 15043666
- [Background] Swithinbank LV, Heron J, von Gontard A, Abrams P. The natural history of daytime urinary incontinence in children: a large British cohort. Acta Paediatr. 2010 Jul;99(7):1031-6. doi: 10.1111/j.1651-2227.2010.01739.x. Epub 2010 Feb 25. PMID 20199496
- [Background] Xing D, Wang YH, Wen YB, Li Q, Feng JJ, Wu JW, Jia ZM, Yang J, Sihoe JD, Song CP, Hu HJ, Franco I, Wen JG. Prevalence and risk factors of overactive bladder in Chinese children: A population-based study. Neurourol Urodyn. 2020 Feb;39(2):688-694. doi: 10.1002/nau.24251. Epub 2019 Dec 5. PMID 31804751
- [Background] Chung JM, Lee SD, Kang DI, Kwon DD, Kim KS, Kim SY, Kim HG, Moon du G, Park KH, Park YH, Pai KS, Suh HJ, Lee JW, Cho WY, Ha TS, Han SW; Korean Enuresis Association. Prevalence and associated factors of overactive bladder in Korean children 5-13 years old: a nationwide multicenter study. Urology. 2009 Jan;73(1):63-7; discussion 68-9. doi: 10.1016/j.urology.2008.06.063. Epub 2008 Sep 30. PMID 18829077
- [Background] Franco I. Overactive bladder in children. Nat Rev Urol. 2016 Sep;13(9):520-32. doi: 10.1038/nrurol.2016.152. Epub 2016 Aug 17. PMID 27530266
- [Background] Fowler CJ, Griffiths D, de Groat WC. The neural control of micturition. Nat Rev Neurosci. 2008 Jun;9(6):453-66. doi: 10.1038/nrn2401. PMID 18490916
- [Background] Griffiths D, Tadic SD. Bladder control, urgency, and urge incontinence: evidence from functional brain imaging. Neurourol Urodyn. 2008;27(6):466-74. doi: 10.1002/nau.20549. PMID 18092336
- [Background] Griffiths D, Tadic SD, Schaefer W, Resnick NM. Cerebral control of the bladder in normal and urge-incontinent women. Neuroimage. 2007 Aug 1;37(1):1-7. doi: 10.1016/j.neuroimage.2007.04.061. Epub 2007 May 18. PMID 17574871
- [Background] Weissbart SJ, Bhavsar R, Rao H, Wein AJ, Detre JA, Arya LA, Smith AL. Specific Changes in Brain Activity during Urgency in Women with Overactive Bladder after Successful Sacral Neuromodulation: A Functional Magnetic Resonance Imaging Study. J Urol. 2018 Aug;200(2):382-388. doi: 10.1016/j.juro.2018.03.129. Epub 2018 Apr 6. PMID 29630979
- [Background] Zuo L, Chen J, Wang S, Zhou Y, Wang B, Gu H. Intra- and inter-resting-state networks abnormalities in overactive bladder syndrome patients: an independent component analysis of resting-state fMRI. World J Urol. 2020 Apr;38(4):1027-1034. doi: 10.1007/s00345-019-02838-z. Epub 2019 Jun 6. PMID 31172280